CLINICAL TRIAL: NCT04996433
Title: Cognitive Behavioral Analysis System of Psychotherapy (CBASP) vs. Behavioral Activation (BA) in Persistently Depressed Treatment-resistant Inpatients: Efficacy, Moderators, and Mediators of Change
Brief Title: A Comparison of Two Psychotherapy Programs in Persistently Depressed Treatment-Resistant Inpatients
Acronym: ChangePDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Greifswald (Other)
Collaborators: German Research Foundation (Other); University of Kassel (Other); University Medicine Greifswald (Other); Charite University, Berlin, Germany (Other); Hannover Medical School (Other); University Hospital Lübeck (Other); Philipps University Marburg (Other); Ludwig-Maximilians - University of Munich (Other); University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BR 4262/6-1
Record Dates: First submitted 2021-06-27; First posted 2021-08-09 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Persistent Depressive Disorder; Treatment-resistant Depression
Keywords: Psychotherapy; Depression; Inpatient Treatment; Childhood Maltreatment; Epigenetic; Moderator; Mediator; Efficacy
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression | interventions — Antidepressive Agents

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, evaluator-blinded, parallel-group, randomized controlled intervention trial with an active control condition
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of interventions, blinding of patients/therapists concerning the treatment program is impossible, but all assessments as well as data analysis will be blinded to treatment allocation. Notably, patients are blinded to the study hypothesis by the Informed Consent process, as patients are told in the patient information and educational discussions about the study that they will in any case receive one of two different scientifically based psychotherapy programs, although it is unclear which of the two programs is more effective. Similarly, the members of the treatment teams of each study ward are not informed about the study hypothesis; however, they are informed that it has not yet been scientifically clarified which therapy is more effective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Analysis System of Psychotherapy (CBASP) (Experimental): Cognitive Behavioral Analysis System of Psychotherapy (CBASP) as acute treatment (5 wk. inpatient and 5 wk. either inpatient or dayclinic) followed by continuation treatment (6 wk. outpatient group therapy).
  Interventions: Behavioral: inpatient CBASP individual therapy; Behavioral: inpatient CBASP group therapy; Behavioral: inpatient CBASP nurse contact; Behavioral: inpatient CBASP exercise therapy; Behavioral: outpatient CBASP group therapy; Drug: algorithm-based study medication
- Behavioral Activation (BA) (Active Comparator): Behavioral Activation (BA) as acute treatment (5 wk. inpatient and 5 wk. either inpatient or dayclinic) followed by continuation treatment (6 wk. outpatient group therapy).
  Interventions: Behavioral: inpatient BA individual therapy; Behavioral: inpatient BA group therapy; Behavioral: inpatient BA nurse contact; Behavioral: inpatient BA exercise therapy; Behavioral: outpatient BA group therapy; Drug: algorithm-based study medication

INTERVENTIONS:
Behavioral: inpatient CBASP individual therapy — During the 5-week inpatient phase I and the 5-week inpatient phase II / dayclinic treatment all patients in this arm will receive 2 individual CBASP therapy sessions (duration: 50 min per session).
  Other Names: Cognitive Behavioral Analysis System of Psychotherapy - inpatient individual therapy
  Arms: Cognitive Behavioral Analysis System of Psychotherapy (CBASP)
Behavioral: inpatient CBASP group therapy — During the 5-week inpatient phase I and the 5-week inpatient phase II / dayclinic treatment all patients in this arm will receive 2 CBASP group therapy sessions (duration: 100 min per session).
  Other Names: Cognitive Behavioral Analysis System of Psychotherapy - inpatient group therapy
  Arms: Cognitive Behavioral Analysis System of Psychotherapy (CBASP)
Behavioral: inpatient CBASP nurse contact — During the 5-week inpatient phase I and the 5-week inpatient phase II / dayclinic treatment all patients in this arm will receive 1 CBASP nurse contact (duration: 30 min per session).
  Other Names: Cognitive Behavioral Analysis System of Psychotherapy - inpatient nurse contact
  Arms: Cognitive Behavioral Analysis System of Psychotherapy (CBASP)
Behavioral: inpatient CBASP exercise therapy — During the 5-week inpatient phase I and the 5-week inpatient phase II / dayclinic treatment all patients in this arm will receive 1 CBASP exercise therapy (duration: 75 min per session).
  Other Names: Cognitive Behavioral Analysis System of Psychotherapy - inpatient exercise therapy
  Arms: Cognitive Behavioral Analysis System of Psychotherapy (CBASP)
Behavioral: outpatient CBASP group therapy — During the 6-week outpatient treatment all patients in this arm will receive 1 CBASP group therapy session (duration: 100 min per session).
  Other Names: Cognitive Behavioral Analysis System of Psychotherapy - outpatient group therapy
  Arms: Cognitive Behavioral Analysis System of Psychotherapy (CBASP)
Behavioral: inpatient BA individual therapy — During the 5-week inpatient phase I and the 5-week inpatient phase II / dayclinic treatment all patients in this arm will receive 2 individual BA therapy sessions (duration: 50 min per session).
  Other Names: Behavioral Activation - inpatient individual therapy
  Arms: Behavioral Activation (BA)
Behavioral: inpatient BA group therapy — During the 5-week inpatient phase I and the 5-week inpatient phase II / dayclinic treatment all patients in this arm will receive 2 BA group therapy sessions (duration: 100 min per session).
  Other Names: Behavioral Activation - inpatient group therapy
  Arms: Behavioral Activation (BA)
Behavioral: inpatient BA nurse contact — During the 5-week inpatient phase I and the 5-week inpatient phase II / dayclinic treatment all patients in this arm will receive 1 BA nurse contact (duration: 30 min per session)
  Other Names: Behavioral Activation - inpatient nurse contact
  Arms: Behavioral Activation (BA)
Behavioral: inpatient BA exercise therapy — During the 5-week inpatient phase I and the 5-week inpatient phase II / dayclinic treatment all patients in this arm will receive 1 BA exercise therapy (duration: 75 min per session).
  Other Names: Behavioral Activation - inpatient exercise therapy
  Arms: Behavioral Activation (BA)
Behavioral: outpatient BA group therapy — During the 6-week outpatient treatment all patients in this arm will receive 1 BA group therapy session (duration: 100 min per session).
  Other Names: Behavioral Activation - outpatient group therapy
  Arms: Behavioral Activation (BA)
Drug: algorithm-based study medication — All patients will receive an optimized, algorithm-based antidepressant medication following the current S3-Guidelines on Unipolar Depression. In case of nonresponse:
  * 1st line dose escalation (if appropriate)
  * 2nd line lithium augmentation
  * 3rd line augmentation with 2nd generation antipsychotics or evidence-based combinations of antidepressants
  * 4th line change of antidepressant.
  Other Names: antidepressant medication

SUMMARY:
The purpose of this study is to compare the Cognitive Behavioral Analysis System of Psychotherapy (CBASP) conducted over 16 weeks (acute and continuation treatment) with Behavioral Activation (BA; same dose and duration) in persistently depressed treatment-resistant inpatients regarding efficacy, moderators and mediators of change.

DETAILED DESCRIPTION:
About half of all psychiatric inpatients with depression suffer from persistent depressive disorder (PDD). Given their high degree of treatment-resistance (TR), comorbidity, suicidality, and hospitalization rates, this patient group appears to be particularly difficult to treat and, from a health economic perspective, constitutes a major challenge. The Cognitive Behavioral Analysis System of Psychotherapy (CBASP) is the only psychotherapy specifically tailored for PDD developed. Originally developed as an outpatient treatment by James P. McCullough, CBASP has been modified for the severely ill PDD patients with TR as a multimodal inpatient concept. Pilot studies indicate very good feasibility and promising outcome. Therefore, a randomized controlled trial is now mandatory for testing the superiority of the inpatient CBASP program vs. the evidence-based Cognitive Behavioral Therapy (CBT), the 'gold standard' in depression treatment. Behavioral Activation (BA) was chosen as the control intervention because BA, as a specific variant of CBT, is at least as effective as standard CBT in severely depressed patients while being easier to train and implement in inpatient settings. Both therapies will be applied as a treatment-phase program (5-week inpatient and dayclinic acute treatment followed by 6-week outpatient continuation group-treatment) in combination with standardized and guideline-based pharmacotherapy. The proposed prospective, multi-center, randomized study with 396 PDD patients with TR will therefore address the primary research question: Is the CBASP program more effective than the BA program in this patient group? The primary hypothesis is that after 16 weeks of treatment, CBASP will show a significant superiority over BA in reducing depressive symptoms. In addition, the important psychotherapy research question: what works for whom and why? will be addressed.

Moderator analyses will examine whether childhood maltreatment and methylation of exon IV of the BDNF gene have an impact on the differential efficacy of the treatments. Regarding mediator analyses, it will be examined whether symptom improvements can be explained by an amelioration of interpersonal problems in CBASP and an increase of activity levels in BA. A follow-up survey 48 weeks after the end of the interventions will provide valuable results regarding the long-term outcome of the treatments. Finally, the health economic potential of the interventions will be investigated through cost-benefit analyses in order to provide important information on the cost-effectiveness of implementation in routine care for health policy. Thus, the results of this study will have the potential to relieve the burden of this very serious and cost-intensive disorder while improving human health. In addition, moderator and mediator analyses may guide personalized treatment and enable therapists to more specifically address psychotherapeutic needs of individual PDD patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-5 diagnosis of PDD (300.4, 296.2x, 296.3x)
* Total Hamilton Depression Rating Scale (HDRS-24) Score ≥ 20
* Treatment-resistance (TR) (defined as a level of 3 or higher on the Antidepressant Treatment History Form: Short Form (ATHF-SF) or medication intolerance or one psychotherapy at least 25 sessions by a certified therapist in the current episode)
* Sufficient knowledge of the German language
* Written informed consent

Exclusion Criteria:

* Bipolar I or II disorder
* Active substance use disorders (abstinence shorter than 6 months)
* Schizophrenia spectrum and other psychotic disorders
* Antisocial personality disorder
* Acute suicidality
* Previous CBASP or BA treatment within the last year
* Inability to tolerate CBASP or BA (e.g., organic brain disorders, severe cognitive deficits)
* Inability to participate in dayclinic or outpatient continuation treatment

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS-24), 24-item version | 16 weeks
  The change in HDRS-24 item score after 16 weeks will be the primary endpoint. The HRSD-24 is a semi-structured interview which is used to measure the severity of all symptom domains of depression as described by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) over a period of the last 7 days. It shows good psychometric properties. The HRSD-24 will be conducted by blind study raters at every time point. Raters evaluate symptom severity on a scale from 0 to 2 or 0 - 3 or 0 - 4 for each item, with higher number indicating higher symptom severity. The total score ranges from 0 to 75 with higher values indicating higher depression severity.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS-24), 24-item version | baseline, weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 64
  The HDRS-24 is a semi-structured interview which is used to measure the severity of all symptom domains of depression as described by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) over a period of the last 7 days. It shows good psychometric properties. The HDRS-24 will be conducted by blind study raters at every time point. Raters evaluate symptom severity on a scale from 0 to 2 or 0 - 3 or 0 - 4 for each item, with higher number indicating higher symptom severity. The total score ranges from 0 to 75 with higher values indicating higher depression severity.
Inventory of Depressive Symptomatology, Self-Report (IDS-SR) | baseline, weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, 32, 40, 48, 56, 64
  The IDS-SR is a self-reported measure of depressive symptoms and used to detect change in self-rated depression severity. It shows good psychometric properties. Each item is rated from 0 to 3 by the patient, and all values are added up to an overall score. Total score ranges from 0 to 78, with higher values indicating a higher depression severity.
Brief Symptom Inventory (BSI) | baseline, weeks 1, 5, 10, 16, 64
  The BSI is a multi-dimensional self-reported measure with a total of nine scales assessing the subjective impairment by physical and psychological symptoms. Each item is rated on a scale from 0 to 5 by the patient and are added up and t-transformed to three global indices: Global Severity Index, Positive Symptom Distress Index, Positive Symptom Total. T-Scores range from 0 to 100, with higher values indicating a higher subjective impairment.
Global Assessment of Functioning (GAF) | baseline, weeks 1, 5, 10, 16, 64
  The GAF is a diagnostic measure used to assess social, occupational and psychological functioning according to DSM-IV. The score ranges from 0 to 100 with a total of ten levels of functioning and is determined by a clinical rater. Higher scores indicate a higher level of functioning and therefore a better outcome.
World Health Organization Quality of Life (WHOQoL-BREF) | baseline, weeks 1, 5, 10, 16, 64
  The WHOQoL-BREF is a self-reporting measure regarding the subjective quality of life. Four broad domains of quality of life are rated by the patient on a five point scale and a mean score for each domain is calculated. Scores range between 4 and 20, with a higher score indicating a higher quality of life and therefore a better outcome.
Response | baseline, weeks 1, 5, 10, 16, 64
  Response (50% decrease on HDRS-24 score)
Remission | baseline, weeks 1, 5, 10, 16, 64
  Remission (HDRS-24 score of 10 or less)
Relapse rates | 16, 64
  Relapse rates (rehospitalization, increase of HDRS-24 of equal or greater than 10 or current HDRS-24 score of equal or greater than 18 points) are measured.
Cost interview | baseline, weeks 16 and 64
  The cost interview assesses direct medical and non-medical costs and indirect costs due to mental disorders versus physical illnesses.

OTHER OUTCOMES:
Childhood Trauma Questionnaire (CTQ) | Baseline
  Childhood maltreatment by the definition of the World Health Organization (WHO) is assessed as a main moderator at baseline. The CTQ measures self-reported childhood trauma on five subscales. Responses are measured on a five point scale, and each subscale score has a range from 5 to 25 points. Higher scores indicate a higher severity in childhood trauma and therefore a worse outcome.
Brain-derived neurotrophic factor (BDNF) | Baseline
  Brain-derived neurotrophic factor (BDNF) methylation as a main moderator.
Inventory of Interpersonal Problems-revised (IIP-32-R) | Baseline, weeks 1, 2, 4, 6, 8, 10, 12, 14, 16 and 64
  The IIP-32-R is a self-reported questionnaire that assesses the severity of interpersonal problems on eight scales based on the two-dimensional interpersonal circumplex model as a main mediator. The items are rated on a five-point scale by the patients. A mean score is calculated, ranging from 0 to 4. A higher score indicates a higher severity of interpersonal problems and therefore a worse outcome.
Behavioral Activation Depression Scale (BADS) | Baseline, weeks 1, 2, 4, 6, 8, 10, 12, 14, 16 and 64
  This self-report is designed to measure weekly changes in avoidance and activation during treatment with Behavioral Activation for depression. The BADS consists of 25 questions on four subscales, each rated on a seven point scale ranging from 0 to 6. The subscales are activation, avoidance/rumination, work/school impairment, and social impairment. A higher total score represents a higher level of activation and therefore a better outcome, while a high score in the subscale social impairment indicates a higher level of impairment and therefore a worse outcome. Scores range from 0 to 150.
Step counts | Baseline, weeks 1, 2, 4, 6, 8, 10, 12, 14, 16 and 64
  Actimeter-measured step-counts as a main mediator.

CONTACTS AND LOCATIONS:
Overall Officials: Eva-Lotta Brakemeier, Prof. Dr., Principal Investigator — University Greifswald
Locations (6):
- Germany (6):
  - Charité, University Medicine Berlin, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Universität zu Lübeck, Lübeck
  - Universitätsklinikum Marburg, Marburg
  - Klinikum der Universität München, München
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the Open Science specifications of the German Psychological Association (DGPS), anonymized data will be made available to the public via the Open Data portal of the Open Science Foundation (www.osf.io). The data will be stored when data collection is completed, but not before 01.01.2028. This step allows third parties to reproduce the analyses reported in scientific publications and to perform ad hoc analyses. The data is permanently stored on servers located in Germany. As soon as they are uploaded and published, these anonymized data cannot be deleted and are therefore also excluded from the deletion of the data in case of revocation of the study participation.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: We will make the outcome data and then the covariate data freely available after our respective publications, but not before 01.01.2028.
Access Criteria: data will be shared with the public; data will be made available for all what types of analyses; the mechanism by which the data will be made available will be determined soon.

REFERENCES:
- [Background] Bernstein DP, Fink LA. CTQ: Childhood Trauma Questionaire: A retrospective self-report.1998; TX: Psychological Corp.
- [Background] Brakemeier EL, Dobias J, Hertel J, Bohus M, Limberger MF, Schramm E, Radtke M, Frank P, Padberg F, Sabass L, Jobst A, Jacob GA, Struck N, Zimmermann J, Normann C. Childhood Maltreatment in Women with Borderline Personality Disorder, Chronic Depression, and Episodic Depression, and in Healthy Controls. Psychother Psychosom. 2018;87(1):49-51. doi: 10.1159/000484481. Epub 2018 Jan 6. No abstract available. PMID 29306947
- [Background] Brakemeier EL, Engel V, Schramm E, Zobel I, Schmidt T, Hautzinger M, Berger M, Normann C. Feasibility and outcome of cognitive behavioral analysis system of psychotherapy (CBASP) for chronically depressed inpatients: a pilot study. Psychother Psychosom. 2011;80(3):191-4. doi: 10.1159/000320779. Epub 2011 Mar 10. No abstract available. PMID 21389759
- [Background] Brakemeier EL, Normann C. Praxisbuch CBASP: Behandlung chronischer Depression; mit Online-Materialien (1. Aufl). 2012. Weinheim: Beltz.
- [Background] Brakemeier EL, Guhn A, Normann C. Praxisbuch CBASP: Behandlung chronischer Depression und Modifikationen für weitere interpersonelle Störungen; mit E-Book inside und Arbeitsmaterial; (2., überarbeitete und erweiterte Auflage). 2021; Weinheim: Beltz.
- [Background] Brakemeier EL, Radtke M, Engel V, Zimmermann J, Tuschen-Caffier B, Hautzinger M, Schramm E, Berger M, Normann C. Overcoming treatment resistance in chronic depression: a pilot study on outcome and feasibility of the cognitive behavioral analysis system of psychotherapy as an inpatient treatment program. Psychother Psychosom. 2015;84(1):51-6. doi: 10.1159/000369586. Epub 2014 Dec 24. PMID 25547778
- [Background] Bschor T, Bauer M, Adli M. Chronic and treatment resistant depression: diagnosis and stepwise therapy. Dtsch Arztebl Int. 2014 Nov 7;111(45):766-75; quiz 775. doi: 10.3238/arztebl.2014.0766. PMID 25467053
- [Background] Cuijpers P, van Straten A, Warmerdam L. Behavioral activation treatments of depression: a meta-analysis. Clin Psychol Rev. 2007 Apr;27(3):318-26. doi: 10.1016/j.cpr.2006.11.001. Epub 2006 Dec 19. PMID 17184887
- [Background] DGPPN, BÄK, KBV, AWMF. S3-Leitlinie/Nationale Versorgungsleitlinie Unipolare Depression- Langfassung: Bd. Version 5 (2. Aufl.). 2015; Springer.
- [Background] Dimidjian S, Hollon SD, Dobson KS, Schmaling KB, Kohlenberg RJ, Addis ME, Gallop R, McGlinchey JB, Markley DK, Gollan JK, Atkins DC, Dunner DL, Jacobson NS. Randomized trial of behavioral activation, cognitive therapy, and antidepressant medication in the acute treatment of adults with major depression. J Consult Clin Psychol. 2006 Aug;74(4):658-70. doi: 10.1037/0022-006X.74.4.658. PMID 16881773
- [Background] Frieling H, Tadic A. Value of genetic and epigenetic testing as biomarkers of response to antidepressant treatment. Int Rev Psychiatry. 2013 Oct;25(5):572-8. doi: 10.3109/09540261.2013.816657. PMID 24151802
- [Background] Guhn A, Kohler S, Brakemeier EL, Sterzer P. Cognitive Behavioral Analysis System of Psychotherapy for inpatients with persistent depressive disorder: a naturalistic trial on a general acute psychiatric unit. Eur Arch Psychiatry Clin Neurosci. 2021 Apr;271(3):495-505. doi: 10.1007/s00406-019-01038-5. Epub 2019 Jul 12. PMID 31300878
- [Background] Harter M, Sitta P, Keller F, Metzger R, Wiegand W, Schell G, Stieglitz RD, Wolfersdorf M, Felsenstein M, Berger M. [Psychiatric-psychotherapeutic inpatient treatment for depression. Process and outcome quality based on a model project in Baden-Wurttemberg]. Nervenarzt. 2004 Nov;75(11):1083-91. doi: 10.1007/s00115-004-1705-8. German. PMID 15197451
- [Background] Holzel L, Wolff Av, Kriston L, Harter M. [Risk factors for non-response in inpatient depression treatment]. Psychiatr Prax. 2010 Jan;37(1):27-33. doi: 10.1055/s-0029-1223348. Epub 2009 Oct 12. German. PMID 19823968
- [Background] Kohler S, Sterzer P, Normann C, Berger M, Brakemeier EL. [Overcoming treatment resistance in chronic depression : The role of inpatient psychotherapy]. Nervenarzt. 2016 Jul;87(7):701-7. doi: 10.1007/s00115-015-0034-4. German. PMID 26610341
- [Background] McCullough JP, Schramm E, Penberthy K. CBASP as a Distinctive Treatment for Persistent Depressive Disorder. 2014; Routledge. https://doi.org/10.4324/9781315743196
- [Background] Nemeroff CB, Heim CM, Thase ME, Klein DN, Rush AJ, Schatzberg AF, Ninan PT, McCullough JP Jr, Weiss PM, Dunner DL, Rothbaum BO, Kornstein S, Keitner G, Keller MB. Differential responses to psychotherapy versus pharmacotherapy in patients with chronic forms of major depression and childhood trauma. Proc Natl Acad Sci U S A. 2003 Nov 25;100(24):14293-6. doi: 10.1073/pnas.2336126100. Epub 2003 Nov 13. PMID 14615578
- [Background] Norcross JC, Wampold BE. Evidence-based therapy relationships: research conclusions and clinical practices. Psychotherapy (Chic). 2011 Mar;48(1):98-102. doi: 10.1037/a0022161. PMID 21401280
- [Background] Richards DA, Ekers D, McMillan D, Taylor RS, Byford S, Warren FC, Barrett B, Farrand PA, Gilbody S, Kuyken W, O'Mahen H, Watkins ER, Wright KA, Hollon SD, Reed N, Rhodes S, Fletcher E, Finning K. Cost and Outcome of Behavioural Activation versus Cognitive Behavioural Therapy for Depression (COBRA): a randomised, controlled, non-inferiority trial. Lancet. 2016 Aug 27;388(10047):871-80. doi: 10.1016/S0140-6736(16)31140-0. Epub 2016 Jul 23. PMID 27461440
- [Background] Sabass L, Padberg F, Normann C, Engel V, Konrad C, Helmle K, Jobst A, Worlitz A, Brakemeier EL. Cognitive Behavioral Analysis System of Psychotherapy as group psychotherapy for chronically depressed inpatients: a naturalistic multicenter feasibility trial. Eur Arch Psychiatry Clin Neurosci. 2018 Dec;268(8):783-796. doi: 10.1007/s00406-017-0843-5. Epub 2017 Sep 27. PMID 28956140
- [Background] Spates CR, Pagoto SL, Kalata A. A qualitative and quantitative review of behavioral activation treatment of major depressive disorder. The Behavior Analyst Today. 2006; 7(4): 508-521. https://doi.org/10.1037/h0100089
- [Background] Shinohara K, Honyashiki M, Imai H, Hunot V, Caldwell DM, Davies P, Moore TH, Furukawa TA, Churchill R. Behavioural therapies versus other psychological therapies for depression. Cochrane Database Syst Rev. 2013 Oct 16;2013(10):CD008696. doi: 10.1002/14651858.CD008696.pub2. PMID 24129886
- [Background] Snarski M, Scogin F, DiNapoli E, Presnell A, McAlpine J, Marcinak J. The effects of behavioral activation therapy with inpatient geriatric psychiatry patients. Behav Ther. 2011 Mar;42(1):100-8. doi: 10.1016/j.beth.2010.05.001. Epub 2010 Nov 20. PMID 21292056
- [Background] Tadic A, Muller-Engling L, Schlicht KF, Kotsiari A, Dreimuller N, Kleimann A, Bleich S, Lieb K, Frieling H. Methylation of the promoter of brain-derived neurotrophic factor exon IV and antidepressant response in major depression. Mol Psychiatry. 2014 Mar;19(3):281-3. doi: 10.1038/mp.2013.58. Epub 2013 May 14. No abstract available. PMID 23670489
- [Background] Struck N, Krug A, Yuksel D, Stein F, Schmitt S, Meller T, Brosch K, Dannlowski U, Nenadic I, Kircher T, Brakemeier EL. Childhood maltreatment and adult mental disorders - the prevalence of different types of maltreatment and associations with age of onset and severity of symptoms. Psychiatry Res. 2020 Nov;293:113398. doi: 10.1016/j.psychres.2020.113398. Epub 2020 Aug 30. PMID 32920524

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT04996433/Prot_SAP_000.pdf